CLINICAL TRIAL: NCT05357586
Title: Serving Those Who Protect the Public: The Pitt Center for Emergency Responder Wellness
Brief Title: The Pitt Center for Emergency Responder Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Eric Meyer, Professor, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21120152
Record Dates: First submitted 2022-04-20; First posted 2022-05-03 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Posttraumatic Stress Disorder; Depression; Anxiety; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: Single group, uncontrolled, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transdiagnostic cognitive behavioral therapy (Experimental): Transdiagnostic cognitive behavioral therapy
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders is a manualized, evidence-based form of cognitive behavioral therapy aimed at targeting emotion regulation processes that underlie common forms of emotional disorders such as anxiety, depression, and commonly co-occurring mental health challenges.

SUMMARY:
Emergency responders protect the public despite occupational hazards that threaten their mental health. The Pitt Center for Emergency Responder Wellness will be a clinical innovation hub that: 1) delivers accessible interventions for promoting mental health and overall wellbeing; 2) trains the next generation of students to provide mental health care for emergency responders; and 3) informs scientific understanding of post-trauma recovery processes. Goals for the seed phase are to establish our team and collect pilot data to demonstrate feasibility and initial clinical impact.

DETAILED DESCRIPTION:
Emergency responders protect the public despite occupational hazards that threaten their mental health. This Center will be a clinical innovation hub that: 1) delivers accessible interventions for promoting mental health and overall wellbeing; 2) trains the next generation of graduate students to provide mental health care for emergency responders; and 3) informs scientific understanding of post-trauma recovery processes. Goals for the seed phase are to establish our team and collect pilot data to demonstrate feasibility and initial clinical impact. In this pilot study, the investigators will demonstrate feasibility by treating 30 eligible emergency responders (up to 60 total participants will be enrolled). The investigators will document treatment acceptability via treatment completion rates. The investigators will document treatment effects by measuring changes in mental health symptoms and quality of life. The investigators will disseminate our findings via conference presentations and manuscripts. The investigators will train graduate students in working with this specialized population.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be age 18 or older.
2. They will be emergency responders defined as fire fighters, law enforcement officers, emergency medical service personnel, emergency room medical providers (physicians, nurses, physician assistants), emergency dispatchers, and emergency response trainees who have completed training experiences in which they encountered emergencies.
3. They must reside in Pennsylvania.

Exclusion Criteria:

1. Are unable or unwilling to complete the study procedures.
2. Receiving another form of therapy our counseling for anxiety, depression, posttraumatic stress, or alcohol use problems. Attendance at self-help programs (e.g., Alcoholics Anonymous) and couples therapy is permitted.
3. Have a history of a psychotic disorder or bipolar disorder.
4. Endorse drug use and symptoms consistent with a non-alcohol substance use disorder except nicotine, caffeine, or cannabis.
5. Are experiencing a current suicidal or homicidal crisis warranting immediate intervention: potential participants may participate later once stabilized.
6. Are currently awaiting the outcome of litigation involving their employment or training as emergency responders or any other reason deemed by the study team to be potentially related to their mental health.
7. Evidence severe organic brain impairment as evidenced by a major apparent disruption of consciousness, cognition, speech, or behavior that would likely interfere with treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline to post-treatment in posttraumatic stress disorder (PTSD) symptom severity using the PTSD Checklist for DSM-5 (PCL-5) | The PCL-5 will be administered at baseline and post-treatment (up to 20 weeks).
  Self-reported posttraumatic stress disorder (PTSD) symptom severity measured using the PCL-5. Scores range from 0-80, with higher scores indicating more severe PTSD symptoms.
Change from baseline to follow-up in posttraumatic stress disorder (PTSD) symptom severity using the PTSD Checklist for DSM-5 (PCL-5) | The PCL-5 will be administered at baseline and follow-up (7 months post-baseline).
  Self-reported posttraumatic stress disorder (PTSD) symptom severity measured using the PCL-5. Scores range from 0-80, with higher scores indicating more severe PTSD symptoms.
Change from baseline to post-treatment in depressive symptom measured using the Patient Health Questionnaire-9 (PHQ-9) | The PHQ-9 will be administered at baseline and post-treatment (up to 20 weeks).
  Self-reported depression symptom severity will be measured using the Patient Health Questionnaire 9 Item-Depression (PHQ-9). Scores range from 0-27, with higher scores indicating greater severity of depression symptoms.
Change from baseline to follow-up in depressive symptoms measured using the Patient Health Questionnaire-9 (PHQ-9) | The PHQ-9 will be administered at baseline and follow-up (7 months post-baseline).
  Self-reported depression symptom severity will be measured using the Patient Health Questionnaire 9 Item-Depression (PHQ-9). Scores range from 0-27, with higher scores indicating greater severity of depression symptoms.
Change from baseline to post-treatment in anxiety symptom severity measured using the Generalized Anxiety Disorder-7 (GAD-7) | The GAD-7 will be administered at baseline and post-treatment (up to 20 weeks).
  Self-reported depression symptom severity measured using the Generalized Anxiety Disorder-7 (GAD-7). Scores range from 0-21 with higher scores indicating greater anxiety symptom severity.
Change from baseline to follow-up in anxiety symptom severity measured using the Generalized Anxiety Disorder-7 (GAD-7) | The GAD-7 will be administered at baseline and follow-up (7 months post-baseline).
  Self-reported depression symptom severity measured using the Generalized Anxiety Disorder-7 (GAD-7). Scores range from 0-21 with higher scores indicating greater anxiety symptom severity.
Change from baseline to post-treatment in alcohol misuse severity measured using the Alcohol Use Disorders Identification Test (AUDIT) | The AUDIT will be administered at baseline and post-treatment (up to 20 weeks).
  Self-reported alcohol misuse measured using the Alcohol Use Disorders Identification Test (AUDIT). Scores range from 0-40 with higher scores indicating greater alcohol misuse.
Change from baseline to follow-up in alcohol misuse severity measured using the Alcohol Use Disorders Identification Test (AUDIT) | The AUDIT will be administered at baseline and follow-up (7 months post-baseline).
  Self-reported alcohol misuse measured using the Alcohol Use Disorders Identification Test (AUDIT). Scores range from 0-40 with higher scores indicating greater alcohol misuse.

SECONDARY OUTCOMES:
Change from baseline to post-treatment in functional impairment measured using the Work and Social Adjustment Scale (WSAS) | The WSAS will be administered at baseline and post-treatment (up to 20 weeks).
  Self-reported functional impairment measured using the Work and Social Adjustment Scale (WSAS). Scores range from 0-8 with higher scores indicating more severe functional impairment.
Change from baseline to follow-up in functional impairment measured using the Work and Social Adjustment Scale (WSAS) | The WSAS will be administered at baseline and follow-up (7 months post-baseline).
  Self-reported functional impairment measured using the Work and Social Adjustment Scale (WSAS). Scores range from 0-8 with higher scores indicating more severe functional impairment.
Change from baseline to post-treatment in quality of life measured using the World Health Organization Quality of Life (WHOQOL-BREF). | The WHOQOL-BREF will be administered at baseline and post-treatment (up to 20 weeks).
  Self-reported quality of life measured using the World Health Organization Quality of Life (WHOQOL-BREF). Scores range from 26 to 130 with higher scores indicating greater quality of life.
Change from baseline to follow-up in quality of life measured using the World Health Organization Quality of Life (WHOQOL-BREF). | The WHOQOL-BREF will be administered at baseline and follow-up (7 months post-baseline).
  Self-reported quality of life measured using the World Health Organization Quality of Life (WHOQOL-BREF). Scores range from 26 to 130 with higher scores indicating greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Meyer, PhD, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers at a future date, either directly or via online research repositories such as Open Science Framework.
  Any necessary transfer agreements will be obtained through the office of research before any data is shared.
Supporting Information: Analytic Code
Time Frame: The data will become available upon the date of the first publication.
Access Criteria: Please contact the Project Director to request data access through a data use agreement.

REFERENCES:
- [Derived] Meyer EC, Roth SG, Coe E, Taylor DJ, Gulliver SB. Pilot outcomes and exploration of treatment mechanisms using a culturally adapted version of the unified protocol for transdiagnostic treatment of emotional disorders to improve mental health symptoms, alcohol misuse, functional outcomes, and sleep quality in emergency responders. Front Health Serv. 2025 Jun 16;5:1452976. doi: 10.3389/frhs.2025.1452976. eCollection 2025. PMID 40589783